CLINICAL TRIAL: NCT04937816
Title: A Meta-Analysis of Amputation Risk in Empagliflozin Studies (1245.25, 1245.110, 1245.121)
Brief Title: This Study Combines Data From 3 Other Studies Testing Empagliflozin in Patients With Diabetes or With Chronic Heart Failure. The Study Looks at the Numbers of Patients Who Had Lower Limb Amputations
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0171
Record Dates: First submitted 2021-06-21; First posted 2021-06-24 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (7):
- EMPA-REG - Placebo: Participants of the EMP-REG OUTCOME study (1245.25) who received placebo.
  Interventions: Drug: Placebo
- EMPA-REG - Empagliflozin low dose: Participants of the EMPA-REG OUTCOME study (1245.25) who received a low dose of empagliflozin once daily (QD).
  Interventions: Drug: Empagliflozin
- EMPA-REG - Empagliflozin high dose: Participants of the EMP-REG OUTCOME study (1245.25) who received a high dose of empagliflozin once daily (QD).
  Interventions: Drug: Empagliflozin
- EMPEROR-Preserved - Empagliflozin: Participants of the EMPEROR-Preserved study (1245.110) who received empagliflozin once daily (QD).
  Interventions: Drug: Empagliflozin
- EMPEROR-Preserved - Placebo: Participants of the EMPEROR-Preserved study (1245.110) who received placebo once daily (QD).
  Interventions: Drug: Placebo
- EMPEROR-Reduced - Empagliflozin: Participants of the EMPEROR-Reduced study (1245.121) who received empagliflozin once daily (QD).
  Interventions: Drug: Empagliflozin
- EMPEROR-Reduced - Placebo: Participants of the EMPEROR-Reduced study (1245.121) who received placebo once daily (QD).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo
  Groups: EMPA-REG - Placebo; EMPEROR-Preserved - Placebo; EMPEROR-Reduced - Placebo
Drug: Empagliflozin — Empagliflozin once daily
  Groups: EMPA-REG - Empagliflozin high dose; EMPA-REG - Empagliflozin low dose; EMPEROR-Preserved - Empagliflozin; EMPEROR-Reduced - Empagliflozin

SUMMARY:
The primary objective of this exploratory meta-analysis is to evaluate the frequencies, incidence rates, and hazard ratios of lower-limb amputation (LLA) events (primary outcome) and of adverse events related to amputation (secondary outcome) in patients treated with empagliflozin compared with placebo in the pooled population of the long-term studies 1245.25, 1245.110, and 1245.121 (SAF-M1), in the pooled population of studies 1245.110 and 1245.121 (SAFM2), and in each of the 3 studies separately.

ELIGIBILITY:
Inclusion Criteria for 1245.25:

* Age ≥18 years, diagnosis of type 2 diabetes mellitus (T2DM)
* Drug-naïve or pretreated with any background therapy
* Glycated haemoglobin (HbA1c) criteria

  * Patients who were drug-naïve: HbA1c of 7 to 10%
  * Patients with background therapy: HbA1c of 7 to 9%
* Body mass index (BMI) ≤45 kg/m2
* With high cardiovascular risk, defined as ≥1 of the following criteria

  * History of myocardial infarction (>2 months prior to enrollment)
  * Multi-vessel coronary artery disease: ≥2 major vessels or left main coronary artery
  * Single-vessel coronary artery disease with no scheduled revascularization/previously unsuccessful revascularization
  * Hospital discharge due to unstable angina pectoris (>2 months prior to enrollment)
  * History of stroke (>2 months prior to enrollment)
  * Peripheral occlusive arterial disease

Inclusion criteria for 1245.110 and 1245.121

* Age ≥18 years (Japan, age ≥20 years)
* Chronic heart failure (HF) new york hear association (NYHA) class II to IV
* Ejection fraction (EF) and N-terminal of the prohormone brain natriuretic peptide (NT-proBNP) criteria

  * 1245.110: preserved EF (Left ventricular ejection fraction (LVEF) >40%) and elevated NT-proBNP (>300 pg/ml; >900 pg/ml for patients with atrial fibrillation)
  * 1245.121: reduced EF (LVEF ≤40%) and elevated NT-proBNP (≥2500 pg/ml if EF 36 to 40%, ≥1000 pg/ml if EF 31 to 35%, ≥600 pg/ml if EF ≤30% or if EF ≤40% with documented hospitalisation for HF within 12 months prior to screening; for patients with atrial fibrillation, double the level of NT-proBNP is applied for each EF category)
* 1245.110 only: structural heart disease within 6 months or documented hospitalisation for HF within 12 months prior to screening
* 1245.121 only: stable dose of medical therapy for HF consistent with local and international cardiology guidelines

Exclusion criteria for 1245.25

* Uncontrolled hyperglycemia: fasting plasma glucose >240 mg/dl
* Severe renal impairment defined as eGFR <30 ml/min by Modification of diet in renal disease (MDRD) formula
* Intake of an investigational drug in another trial within 30 days prior to intake of study medication in this trial, or participating in another trial (involving an investigational drug and/or follow-up)

Exclusion criteria for 1245.110 and 1245.121

* Myocardial infarction, coronary artery bypass graft surgery or other major cardiovascular surgery, stroke or transient ischaemic attack ≤90 days before screening
* Heart transplant recipient, or listed for heart transplant
* Acute decompensated HF
* Systolic blood pressure (SBP) ≥180 mmHg at randomisation
* Symptomatic hypotension and/or SBP <100 mmHg at screening or randomisation
* Impaired renal function defined as Estimated glomerular filtration rate (eGFR) Chronic Kidney Disease Epidemiology Collaboration Equation (based on serum creatinine value) <20 ml/min/1.73 m2 or requiring dialysis at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus and increased cardiovascular risk (1245.25), patients with chronic heart failure with preserved ejection fraction (1245.110), and patients with chronic heart failure with reduced ejection fraction (1245.121), who were either treated with empagliflozin or placebo.
Sampling Method: Non-Probability Sample
Enrollment: 16746 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim, Ingelheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This meta-analysis includes three randomised, placebo-controlled, double-blind, parallel-group and event-driven studies (NCT01131676, NCT03057951, NCT03057977) to evaluate the risk of lower-limb amputation (LLA) in patients treated with empagliflozin compared to placebo in the pooled population (SAF-M1 vs. SAF-M2).
Pre-assignment Details: As this is a meta-analysis of three independent trials, all subjects were screened for eligibility prior to participation of the respective trial.
Groups:
- Trial NCT01131676: Placebo: Oral administration of Placebo matching empagliflozin 10 or 25 milligram (mg) (1 tablet once daily) in patients with type 2 diabetes mellitus (T2DM).
- Trial NCT01131676: Empagliflozin 10 mg: 1 film-coated tablet of 10 mg empagliflozin (BI 10773) was administered orally once daily in patients with T2DM.
- Trial NCT01131676: Empagliflozin 25 mg: 1 film-coated tablet of 25 mg empagliflozin (BI 10773) was administered orally once daily in patients with T2DM.
- Trial NCT03057951: Placebo: 1 film-coated tablet of matching placebo was administered orally once daily in patients with chronic heart failure with preserved ejection fraction (HFpEF).
- Trial NCT03057951: Empagliflozin 10 mg: 1 film-coated tablet of 10 milligram (mg) of empagliflozin (BI 10773) was administered orally once daily in patients with chronic heart failure with preserved ejection fraction (HFpEF).
- Trial NCT03057977: Placebo: 1 film-coated tablet of matching placebo was administered orally once daily in patients with heart failure with reduced ejection fraction (HFrEF).
- Trial NCT03057977: Empagliflozin 10 mg: 1 film-coated tablet of 10 milligram (mg) empagliflozin (BI 10773) was administered orally once daily in patients with heart failure with reduced ejection fraction (HFrEF).
Period: Overall Study
Arm/Group | Trial NCT01131676: Placebo | Trial NCT01131676: Empagliflozin 10 mg | Trial NCT01131676: Empagliflozin 25 mg | Trial NCT03057951: Placebo | Trial NCT03057951: Empagliflozin 10 mg | Trial NCT03057977: Placebo | Trial NCT03057977: Empagliflozin 10 mg
Started (Randomised) | 2337 | 2347 | 2344 | 2991 | 2997 | 1867 | 1863
Treated | 2333 | 2345 | 2342 | 2989 | 2996 | 1863 | 1863
Completed | 1650 | 1790 | 1800 | 2046 | 2051 | 1352 | 1381
Not Completed | 687 | 557 | 544 | 945 | 946 | 515 | 482
Not completed — Study drug stopped, reason missing | 5 | 3 | 4 | 6 | 1 | 0 | 0
Not completed — Other than stated below | 173 | 143 | 125 | 44 | 45 | 28 | 31
Not completed — Patient refusal to continue, not due to AE | 172 | 118 | 122 | 304 | 284 | 124 | 92
Not completed — Lost to Follow-up | 15 | 9 | 6 | 6 | 16 | 11 | 17
Not completed — Protocol Violation | 15 | 15 | 12 | 30 | 24 | 5 | 5
Not completed — Adverse Event | 303 | 267 | 273 | 553 | 575 | 343 | 337
Not completed — Not treated | 4 | 2 | 2 | 2 | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): Patients treated with at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trial NCT01131676: Placebo | Trial NCT01131676: Empagliflozin 10 mg | Trial NCT01131676: Empagliflozin 25 mg | Trial NCT03057951: Placebo | Trial NCT03057951: Empagliflozin 10 mg | Trial NCT03057977: Placebo | Trial NCT03057977: Empagliflozin 10 mg | Total
Number analyzed (Participants) | 2333 | 2345 | 2342 | 2989 | 2996 | 1863 | 1863 | 16731
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (8.8) | 63.0 (8.6) | 63.2 (8.6) | 71.9 (9.6) | 71.8 (9.3) | 66.5 (11.2) | 67.2 (10.8) | 67.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 653 | 692 | 659 | 1336 | 1338 | 453 | 437 | 5568
  Male | 1680 | 1653 | 1683 | 1653 | 1658 | 1410 | 1426 | 11163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 418 | 432 | 415 | 753 | 770 | 613 | 616 | 4017
  Not Hispanic or Latino | 1912 | 1909 | 1926 | 2235 | 2226 | 1175 | 1164 | 12547
  Unknown or Not Reported | 3 | 4 | 1 | 1 | 0 | 75 | 83 | 167
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 20 | 11 | 23 | 104 | 90 | 24 | 15 | 287
  Asian | 511 | 505 | 501 | 411 | 413 | 334 | 337 | 3012
  Native Hawaiian or Other Pacific Islander | 4 | 3 | 3 | 19 | 14 | 6 | 8 | 57
  Black or African American | 120 | 119 | 118 | 125 | 133 | 134 | 123 | 872
  White | 1678 | 1707 | 1696 | 2254 | 2285 | 1301 | 1325 | 12246
  More than one race | 0 | 0 | 0 | 75 | 60 | 33 | 28 | 196
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 1 | 31 | 27 | 61

OUTCOME MEASURES:

1. Secondary Outcome: Incidence Rate of Adverse Events Related to Amputation
Description: Incidence rate of adverse events (AEs) related to amputation. Incidence rate were provided as rate per 100 patients-years (pt-yrs) calculated as the observed number of patients with event divided by observed time-at-risk over all patients.
  Time at risk was derived as followed:
  Patient with event:
  time at risk in days = date of start of first event - treatment start date + 1.
  Patients without event:
  time at risk in days = last date on treatment + 7 days - treatment start date + 1.
  A search with a pre-defined list of MedDRA preferred terms was performed to identify all AEs related to amputation. These AE included vascular disorders, diabetic-foot-related events, wound/infections, nervous system disorders and volume depletion events.
  Abbreviation: pt-yrs = patient-years.
Time Frame: From first to last dose of study medication plus 7 days to account for the residual drug effect, up to 1639 days.
Population: Treated Set: Patients treated with at least 1 dose of study medication. Results are reported by the pooled population (SAF-M1 and SAF-M2) and for each study separately. For trial NCT01131676, 10 mg and 25 mg were combined, as the overall safety profile is similar for empagliflozin 10 mg and 25 mg. This approach was agreed with the European Medicines Agency (EMA).
Measure: Number (95% Confidence Interval); unit: Patients with events per 100 pt-yrs
Groups:
- SAF-M1 Placebo: Safety analysis grouping (SAF)-M1 - Placebo included the pooled population of all three studies. Patients with type 2 diabetes mellitus (T2DM) (NCT01131676), patients with heart failure with preserved ejection fraction (HFpEF) (NCT03057951) and patients with heart failure with reduced ejection fraction (HFrEF) (NCT03057977) treated with placebo. In all three trials, 1 film-coated tablet of placebo matching empagliflozin was administered orally once daily.
- SAF-M1 Empagliflozin: Safety analysis grouping (SAF)-M1 included the pooled population of all three studies. Patients with T2DM (NCT01131676), patients with HFpEF (NCT03057951) and patients with HFrEF (NCT03057977) treated with 10 milligram (mg) or 25 mg empagliflozin.
- SAF-M2 Placebo: SAF-M2 included the pooled population of the 2 chronic heart failure studies (NCT03057951, NCT03057977). Patients with HFpEF and patients with HFrEF treated with placebo. In both trials, 1 film-coated tablet of placebo matching empagliflozin was administered orally once daily.
- SAF-M2 Empagliflozin 10 mg: SAF-M2 included the pooled population of the 2 chronic heart failure studies (NCT03057951, NCT03057977). Patients with HFpEF and patients with HFrEF treated with 10 mg empagliflozin, administered as film-coated tablet orally once daily.
- Trial NCT01131676: Empagliflozin 10 mg or 25 mg: 1 film-coated tablet of 10 mg or 25 mg empagliflozin (BI 10773) was administered orally once daily in patients with T2DM.
Arm/Group | SAF-M1 Placebo | SAF-M1 Empagliflozin | SAF-M2 Placebo | SAF-M2 Empagliflozin 10 mg | Trial NCT01131676: Placebo | Trial NCT01131676: Empagliflozin 10 mg or 25 mg | Trial NCT03057951: Placebo | Trial NCT03057951: Empagliflozin 10 mg | Trial NCT03057977: Placebo | Trial NCT03057977: Empagliflozin 10 mg
Number analyzed (Participants) | 7185 | 9546 | 4852 | 4859 | 2333 | 4687 | 2989 | 2996 | 1863 | 1863
Patients with events per 100 pt-yrs
  Vascular adverse event | 1.48 [1.28 to 1.69] | 1.57 [1.40 to 1.75] | 1.27 [1.03 to 1.54] | 1.21 [0.98 to 1.47] | 1.77 [1.44 to 2.13] | 1.81 [1.57 to 2.06] | 1.21 [0.94 to 1.51] | 1.17 [0.90 to 1.47] | 1.44 [0.98 to 1.97] | 1.33 [0.90 to 1.85]
  Diabetic foot related AE | 0.50 [0.39 to 0.63] | 0.64 [0.53 to 0.76] | 0.32 [0.21 to 0.46] | 0.46 [0.32 to 0.62] | 0.75 [0.54 to 0.99] | 0.76 [0.62 to 0.93] | 0.38 [0.23 to 0.55] | 0.30 [0.18 to 0.46] | 0.18 [0.05 to 0.39] | 0.84 [0.51 to 1.26]
  Infections potentially related to LLA | 2.19 [1.94 to 2.44] | 2.04 [1.85 to 2.25] | 1.85 [1.56 to 2.17] | 1.78 [1.50 to 2.09] | 2.64 [2.23 to 3.09] | 2.22 [1.96 to 2.50] | 1.97 [1.62 to 2.36] | 1.75 [1.42 to 2.11] | 1.57 [1.09 to 2.13] | 1.88 [1.35 to 2.49]
  Wound/infection | 0.86 [0.71 to 1.02] | 0.86 [0.73 to 0.99] | 0.65 [0.49 to 0.84] | 0.46 [0.32 to 0.62] | 1.14 [0.87 to 1.43] | 1.12 [0.94 to 1.32] | 0.61 [0.42 to 0.83] | 0.48 [0.32 to 0.68] | 0.76 [0.44 to 1.16] | 0.40 [0.18 to 0.70]
  Nervous system disorder | 1.54 [1.34 to 1.76] | 1.81 [1.62 to 2.00] | 0.85 [0.66 to 1.07] | 0.92 [0.72 to 1.14] | 2.53 [2.12 to 2.96] | 2.41 [2.14 to 2.70] | 0.92 [0.69 to 1.19] | 0.99 [0.74 to 1.27] | 0.67 [0.37 to 1.05] | 0.75 [0.44 to 1.15]
  Volume depletion | 0.67 [0.54 to 0.81] | 0.65 [0.54 to 0.77] | 0.95 [0.75 to 1.18] | 1.16 [0.94 to 1.41] | 0.28 [0.16 to 0.43] | 0.32 [0.23 to 0.43] | 0.90 [0.67 to 1.17] | 1.16 [0.90 to 1.46] | 1.08 [0.69 to 1.55] | 1.16 [0.76 to 1.64]
Statistical Analysis 1: Comparison: SAF-M1 Placebo vs SAF-M1 Empagliflozin; Time to first vascular AE (SAF-M1); Test type: Other; p = 0.9946, Regression, Cox; Cox regression of time to first vascular AE. Cox regression model with terms for study, baseline diabetes status and treatment; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.83 to 1.20] — Comparison versus Placebo [Treatment/ Placebo]
Statistical Analysis 2: Comparison: SAF-M2 Placebo vs SAF-M2 Empagliflozin 10 mg; Time to first vascular AE (SAF-M2); Test type: Other; p = 0.7474, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.72 to 1.27] — Comparison versus placebo. [Treatment/Placebo]
Statistical Analysis 3: Comparison: Trial NCT01131676: Placebo vs Trial NCT01131676: Empagliflozin 10 mg or 25 mg; Time to first vascular AE (Trial NCT01131676, all empagliflozin (10 and 25 mg vs. Placebo)); Test type: Other; p = 0.7943, Regression, Cox; Cox regression for time to first vascular AE on-treatment. Cox regression model with a term for treatment; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.81 to 1.31] — Comparison vs. Placebo [Treatment / Placebo]
Statistical Analysis 4: Comparison: Trial NCT03057951: Placebo vs Trial NCT03057951: Empagliflozin 10 mg; Time to first vascular AE (Trial NCT03057951); Test type: Other; p = 0.8518, Regression, Cox; Cox regression for time to first vascular AE on-treatment. Cox regression model with terms for baseline diabetes status and treatment; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.69 to 1.36] — Comparison vs. Placebo [Treatment / Placebo]
Statistical Analysis 5: Comparison: Trial NCT03057977: Placebo vs Trial NCT03057977: Empagliflozin 10 mg; Time to first vascular AE (Trial NCT03057977); Test type: Other; p = 0.7660, Regression, Cox; [statistical method as in outcome 1, analysis 4]; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.56 to 1.53] — Comparison vs Placebo [Treatment/Placebo]
Statistical Analysis 6: Comparison: SAF-M1 Placebo vs SAF-M1 Empagliflozin; Time to first diabetic foot related AE (SAF-M1); Test type: Other; p = 0.3612, Regression, Cox; Cox regression of time to first diabetic foot related AE. Cox regression model with terms for study, baseline diabetes status and treatment; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.85 to 1.55] — Comparison versus placebo [Treatment/Placebo]
Statistical Analysis 7: Comparison: SAF-M2 Placebo vs SAF-M2 Empagliflozin 10 mg; Time to first diabetic foot related AE (SAF-M2); Test type: Other; p = 0.1610, Regression, Cox; [statistical method as in outcome 1, analysis 6]; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [0.86 to 2.40] — Comparison versus Placebo [Treatment/Placebo]
Statistical Analysis 8: Comparison: Trial NCT01131676: Placebo vs Trial NCT01131676: Empagliflozin 10 mg or 25 mg; Time to first diabetic foot related AE (Trial NCT01131676, all empagliflozin (10 and 25 mg) vs. Placebo); Test type: Other; p = 0.9128, Regression, Cox; Cox regression for time to first diabetic foot related AE on treatment. Cox regression model with a term for treatment; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.71 to 1.47] — Comparison vs. Placebo [Treatment/Placebo]
Statistical Analysis 9: Comparison: Trial NCT03057951: Placebo vs Trial NCT03057951: Empagliflozin 10 mg; Time to first diabetic foot related AE (Trial NCT03057951); Test type: Other; p = 0.5276, Regression, Cox; Cox regression for time to first diabetic foot related AE. Cox regression model with terms for baseline diabetes status and treatment; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.43 to 1.54] — Comparison vs. Placebo [Treatment/Placebo]
Statistical Analysis 10: Comparison: Trial NCT03057977: Placebo vs Trial NCT03057977: Empagliflozin 10 mg; Time to first diabetic foot related AE (Trial NCT03057977); Test type: Other; p = 0.0048, Regression, Cox; [statistical method as in outcome 1, analysis 9]; Hazard Ratio (HR) = 4.72, 95% CI 2-sided [1.60 to 13.87] — Comparison vs Placebo [Treatment / Placebo]
Statistical Analysis 11: Comparison: SAF-M1 Placebo vs SAF-M1 Empagliflozin; Time to first infections potentially related to LLA's (SAF-M1); Test type: Other; p = 0.1526, Regression, Cox; Cox regression of time to first infections potentially related to LLA's. Cox regression with terms for study, baseline diabetes status and treatment; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.77 to 1.04] — Comparison versus Placebo [Treatment/Placebo]
Statistical Analysis 12: Comparison: SAF-M2 Placebo vs SAF-M2 Empagliflozin 10 mg; Time to first infection potentially related to LLA's (SAF-M2); Test type: Other; p = 0.7430, Regression, Cox; Cox regression of time to first infection potentially related to LLA's. Cox regression with terms for study, baseline diabetes status and treatment; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.76 to 1.21] — Comparison versus Placebo [Treatment/Placebo]
Statistical Analysis 13: Comparison: Trial NCT01131676: Placebo vs Trial NCT01131676: Empagliflozin 10 mg or 25 mg; Time to first infections potentially related to LLA (Trial NCT01131676, all Empagliflozin (10 mg and 25 mg) vs. Placebo); Test type: Other; p = 0.1049, Regression, Cox; Cox regression for infections potentially related to LLA-on treatment. Cox regression model with a term for treatment; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.69 to 1.04] — Comparison vs Placebo [Treatment/Placebo]
Statistical Analysis 14: Comparison: Trial NCT03057951: Placebo vs Trial NCT03057951: Empagliflozin 10 mg; Time to first infections potentially related to LLA (Trial NCT03057951); Test type: Other; p = 0.3950, Regression, Cox; Cox regression for infections potentially related to LLA on treatment. Cox regression model with terms for baseline diabetes status and treatment; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.67 to 1.17] — Comparison vs Placebo [Treatment/Placebo]
Statistical Analysis 15: Comparison: Trial NCT03057977: Placebo vs Trial NCT03057977: Empagliflozin 10 mg; Time to first infections potentially related to LLA (Trial NCT03057977); Test type: Other; p = 0.4429, Regression, Cox; Cox regression for infections potentially related to LLA on-treatment. Cox regression model with terms for baseline diabetes status and treatment; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.76 to 1.87] — Comparison vs Placebo [Treatment/Placebo]
Statistical Analysis 16: Comparison: SAF-M1 Placebo vs SAF-M1 Empagliflozin; Time to first wound/infection (SAF-M1); Test type: Other; p = 0.3396, Regression, Cox; Cox regression of time to first wound infections. Cox regression with terms for study, baseline diabetes status and treatment; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.70 to 1.13] — Comparison versus Placebo [Treatment/Placebo]
Statistical Analysis 17: Comparison: SAF-M2 Placebo vs SAF-M2 Empagliflozin 10 mg; Time to first wound/infection (SAF-M2); Test type: Other; p = 0.1050, Regression, Cox; [statistical method as in outcome 1, analysis 16]; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.46 to 1.08] — Comparison versus Placebo [Treatment/Placebo]
Statistical Analysis 18: Comparison: Trial NCT01131676: Placebo vs Trial NCT01131676: Empagliflozin 10 mg or 25 mg; Time to first wound/infection (Trial NCT01131676, all Empagliflozin (10 mg and 25 mg) vs Placebo); Test type: Other; p = 0.9919, Regression, Cox; Cox regression for time to first wound/infection on-treatment; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.74 to 1.35] — Comparison vs Placebo [Treatment/Placebo]
Statistical Analysis 19: Comparison: Trial NCT03057951: Placebo vs Trial NCT03057951: Empagliflozin 10 mg; Time to first wound/infection (Trial NCT03057951); Test type: Other; p = 0.3634, Regression, Cox; Cox regression for time to first wound/infection on-treatment. Cox regression model with terms for baseline diabetes status and treatment; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.48 to 1.31] — Comparison vs Placebo [Treatment/Placebo]
Statistical Analysis 20: Comparison: Trial NCT03057977: Placebo vs Trial NCT03057977: Empagliflozin 10 mg; Time to first wound/infection (Trial NCT03057977); Test type: Other; p = 0.1177, Regression, Cox; [statistical method as in outcome 1, analysis 19]; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.23 to 1.18] — Comparison vs Placebo [Treatment/Placebo]
Statistical Analysis 21: Comparison: SAF-M1 Placebo vs SAF-M1 Empagliflozin; Time to first nervous system disorder (SAF-M1); Test type: Other; p = 0.9992, Regression, Cox; Cox regression of time to first nervous system disorder. Cox regression with terms for study, baseline diabetes status and treatment; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.84 to 1.19] — Comparison versus Placebo [Treatment/Placebo]
Statistical Analysis 22: Comparison: SAF-M2 Placebo vs SAF-M2 Empagliflozin 10 mg; Time to first nervous system disorder (SAF-M2); Test type: Other; p = 0.6274, Regression, Cox; Cox regression of time to first nervous system disorder. Cox regression model with terms for study, baseline diabetes status and treatment; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.78 to 1.52] — Comparison versus Placebo [Treatment/Placebo]
Statistical Analysis 23: Comparison: Trial NCT01131676: Placebo vs Trial NCT01131676: Empagliflozin 10 mg or 25 mg; Time to first nervous system disorder (Trial NCT01131676, all Empagliflozin (10 mg and 25 mg) vs Placebo); Test type: Other; p = 0.7597, Regression, Cox; Cox regression for time to first nervous system disorder on-treatment. Cox regression model with a term for treatment; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.79 to 1.19] — Comparison vs Placebo [Treatment/Placebo]
Statistical Analysis 24: Comparison: Trial NCT03057951: Placebo vs Trial NCT03057951: Empagliflozin 10 mg; Time to first nervous system disorder (Trial NCT03057951); Test type: Other; p = 0.7067, Regression, Cox; Cox regression for time to first nervous system disorder on-treatment. Cox regression model with terms for baseline diabetes status and treatment; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.74 to 1.57] — Comparison vs Placebo [Treatment/Placebo]
Statistical Analysis 25: Comparison: Trial NCT03057977: Placebo vs Trial NCT03057977: Empagliflozin 10 mg; time to first nervous system disorder (Trial NCT03057977); Test type: Other; p = 0.7404, Regression, Cox; [statistical method as in outcome 1, analysis 24]; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.56 to 2.25] — Comparison vs Placebo [Treatment/Placebo]
Statistical Analysis 26: Comparison: SAF-M1 Placebo vs SAF-M1 Empagliflozin; Time to first volume depletion AE (SAF-M1); Test type: Other; p = 0.1765, Regression, Cox; Cox regression of time to first volume depletion AE. Cox regression model with terms for study, baseline diabetes status and treatment; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.92 to 1.58] — Comparison versus Placebo [Treatment/Placebo]
Statistical Analysis 27: Comparison: SAF-M2 Placebo vs SAF-M2 Empagliflozin 10 mg; Time to first volume depletion AE (SAF-M2); Test type: Other; p = 0.1978, Regression, Cox; Cox regression of time to first volume depletion AE. Cox regression with terms for study, baseline diabetes status and treatment; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.90 to 1.66] — Comparison versus Placebo [Treatment/Placebo]
Statistical Analysis 28: Comparison: Trial NCT01131676: Placebo vs Trial NCT01131676: Empagliflozin 10 mg or 25 mg; Time to first volume depletion (Trial NCT01131676, all Empagliflozin (10 mg and 25 mg) vs Placebo); Test type: Other; p = 0.6561, Regression, Cox; Cox regression for time to first volume depletion on-treatment. Cox regression model with a term for treatment; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.64 to 2.05] — Comparison vs Placebo [Treatment/Placebo]
Statistical Analysis 29: Comparison: Trial NCT03057951: Placebo vs Trial NCT03057951: Empagliflozin 10 mg; Time to first volume depletion (Trial NCT03057951); Test type: Other; p = 0.1699, Regression, Cox; Cox regression for time to first volume depletion on-treatment. Cox regression model with terms for baseline diabetes status and treatment; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.90 to 1.87] — Comparison vs Placebo [Treatment/Placebo]
Statistical Analysis 30: Comparison: Trial NCT03057977: Placebo vs Trial NCT03057977: Empagliflozin 10 mg; Time to first volume depletion (Trial NCT03057977); Test type: Other; p = 0.7944, Regression, Cox; [statistical method as in outcome 1, analysis 29]; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.62 to 1.87] — Comparison vs Placebo [Treatment/Placebo]

2. Primary Outcome: Incidence Rate of Lower Limb Amputation (LLA)
Description: Incidence rate of lower limb amputation (LLA). Incidence rate were provided as rate per 100 patients-years (pt-yrs) calculated as the observed number of patients with event divided by observed time-at-risk over all patients.
  Time at risk was derived as followed:
  Patient with event:
  time at risk in days = date of start of first event - treatment start date + 1.
  Patients without event:
  time at risk in days = last date on treatment + 7 days - treatment start date + 1.
  Abbreviation: pt-yrs = patient-years.
Time Frame: From first to last dose of study medication plus 7 days to account for the residual drug effect, up to 1639 days.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Patients with events per 100pt-yrs
Arm/Group | SAF-M1 Placebo | SAF-M1 Empagliflozin | SAF-M2 Placebo | SAF-M2 Empagliflozin 10 mg | Trial NCT01131676: Placebo | Trial NCT01131676: Empagliflozin 10 mg or 25 mg | Trial NCT03057951: Placebo | Trial NCT03057951: Empagliflozin 10 mg | Trial NCT03057977: Placebo | Trial NCT03057977: Empagliflozin 10 mg
Number analyzed (Participants) | 7185 | 9546 | 4852 | 4859 | 2333 | 4687 | 2989 | 2996 | 1863 | 1863
Patients with events per 100pt-yrs | 0.40 [0.30 to 0.52] | 0.48 [0.39 to 0.58] | 0.27 [0.17 to 0.39] | 0.23 [0.13 to 0.34] | 0.59 [0.41 to 0.81] | 0.64 [0.51 to 0.79] | 0.27 [0.15 to 0.42] | 0.20 [0.10 to 0.33] | 0.27 [0.10 to 0.52] | 0.31 [0.12 to 0.58]
Statistical Analysis 1: Comparison: SAF-M1 Placebo vs SAF-M1 Empagliflozin; Test type: Other; p = 0.9276, Regression, Cox; Cox regression model with terms for study, baseline diabetes status and treatment; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.73 to 1.42] — Comparison versus placebo [Treatment/Placebo]
Statistical Analysis 2: Comparison: SAF-M2 Placebo vs SAF-M2 Empagliflozin 10 mg; Test type: Other; p = 0.6205, Regression, Cox; Cox regression model with terms for study, baseline diabetes status and treatment; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.45 to 1.60] — Comparison versus placebo [Treatment/Placebo]
Statistical Analysis 3: Comparison: Trial NCT01131676: Placebo vs Trial NCT01131676: Empagliflozin 10 mg or 25 mg; Empagliflozin (10 mg + 25 mg) versus Placebo; Test type: Other; p = 0.6768, Regression, Cox; Cox regression model with terms for treatment; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.73 to 1.63] — Comparison vs Placebo [Treatment/Placebo]
Statistical Analysis 4: Comparison: Trial NCT03057951: Placebo vs Trial NCT03057951: Empagliflozin 10 mg; Test type: Other; p = 0.4294, Regression, Cox; Cox regression model with terms for baseline diabetes status and treatment; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.34 to 1.59] — Comparison versus Placebo [Treatment /Placebo]
Statistical Analysis 5: Comparison: Trial NCT03057977: Placebo vs Trial NCT03057977: Empagliflozin 10 mg; Test type: Other; p = 0.7826, Regression, Cox; Cox regression model with terms for baseline diabetes status and treatment; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.39 to 3.47] — Comparison versus Placebo [Treatment /Placebo]

ADVERSE EVENTS:
Description: As this is a meta-analysis adverse events were not planned to be collected and reported. Adverse events of each study (NCT01131676, NCT03057951, NCT03057977) included in this meta-analysis have already been disclosed.
Groups:
- SAF-M1 Empagliflozin 10 mg: Safety analysis grouping (SAF)-M1 Empagliflozin 10 mg included the pooled population of all three studies. Patients with T2DM (NCT01131676), patients with HFpEF (NCT03057951) and patients with HFrEF (NCT03057977) treated with 10 milligram (mg) empagliflozin. In all three trials, a film-coated tablet of 10 mg Empagliflozin was administered orally once daily.
- SAF-M1 Empagliflozin 25 mg: Safety analysis grouping (SAF)-M1 Empagliflozin 25 mg included the pooled population of trial NCT01131676. Patients were administered one film-coated tablet of 25 milligram (mg) empagliflozin orally once daily.
Arm/Group | SAF-M1 Placebo | SAF-M1 Empagliflozin 10 mg | SAF-M1 Empagliflozin 25 mg | SAF-M2 Placebo | SAF-M2 Empagliflozin 10 mg | Trial NCT01131676: Placebo | Trial NCT01131676: Empagliflozin 10 mg | Trial NCT01131676: Empagliflozin 25 mg | Trial NCT03057977: Placebo | Trial NCT03057977: Empagliflozin 10 mg | Trial NCT03057951: Placebo | Trial NCT03057951: Empagliflozin 10 mg
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
For study NCT01131676, events leading to LLA were not prespecified but were identified during unblinded medical review of data. Also, since both empagliflozin arms (10 and 25 mg) of study NCT01131676 were combined for the pooled SAF-M1 analysis, this led not only to a different sample size, but also to different patient populations for placebo and empagliflozin, respectively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT04937816/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT04937816/SAP_001.pdf